CLINICAL TRIAL: NCT07350746
Title: A Comparison of Outcome of Pulpotomy on Immature Permanent Molars Between Different Calcium Silicate-based Materials : a 12 Months Clinical Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint-Joseph University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USJ- CER-2025-289
Record Dates: First submitted 2025-11-29; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Pain; Lesions
MeSH Terms: conditions — Pain | interventions — International Normalized Ratio

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neo PUTTY (Nusmile Inc, Houston, TX; USA) (Experimental): premixed bioactive bioceramic composed of an inorganic powder containing tricalcium and dicalcium silicate in a water-free organic liquid.
  Interventions: Device: Neo PUTTY (Nusmile Inc, Houston, TX; USA)
- Total Fill® BC UNIVERSAL RRM™ (FKG Dentaire, Switzerland) (Active Comparator): premixed bioceramic material composed of calcium aluminosilicate paste designed for permanent root canal repair and surgical applications.
  Interventions: Device: Total Fill® BC UNIVERSAL RRM™ (FKG Dentaire, Switzerland)
- Bio-C® Repair (BCR; Angelus, Londrina, Brazil) (Active Comparator): new ready-to-use bioceramic repair material. Bio-C has indications similar to MTA and is composed of calcium silicates [tricalcium silicate, dicalcium silicate], tricalcium aluminate, calcium oxide (for the release of calcium ions), and zirconium oxide as a radioopacifier.
  Interventions: Device: Bio-C® Repair (BCR; Angelus, Londrina, Brazil)

INTERVENTIONS:
Device: Bio-C® Repair (BCR; Angelus, Londrina, Brazil) — To the best of our knowledge, no study has yet compared these three biomaterials in the treatment of permanent molars with incomplete root development.
  Arms: Bio-C® Repair (BCR; Angelus, Londrina, Brazil)
Device: Total Fill® BC UNIVERSAL RRM™ (FKG Dentaire, Switzerland) — To the best of our knowledge, no study has yet compared these three biomaterials in the treatment of permanent molars with incomplete root development.
  Arms: Total Fill® BC UNIVERSAL RRM™ (FKG Dentaire, Switzerland)
Device: Neo PUTTY (Nusmile Inc, Houston, TX; USA) — To the best of our knowledge, no study has yet compared these three biomaterials in the treatment of permanent molars with incomplete root development.
  Arms: Neo PUTTY (Nusmile Inc, Houston, TX; USA)

SUMMARY:
Preservation of pulp vitality through vital pulp therapy (VPT) has emerged in contemporary endodontics, particularly for immature permanent teeth. In cases of irreversible pulpitis, recent literature suggests that clinical symptoms do not always correlate with histopathological findings, supporting the use of conservative approaches such as full pulpotomy. This is especially relevant in young patients where continued root development and apical closure are critical for long-term tooth integrity and functionality. Immature teeth, due to their high cellularity and vascularity, exhibit a greater regenerative capacity, making them indicated for biologically based treatments.

Among the materials used for VPT, calcium silicate-based cements (CSCs) have demonstrated good biological and physicochemical properties, including high biocompatibility, antimicrobial effects, alkaline pH, and sustained release of calcium ions that stimulate biomineralization. Mineral Trioxide Aggregate (MTA) has long been considered the gold standard; however, it is associated with several clinical limitations such as extended setting time, complex handling, and potential tooth discoloration. To address these drawbacks, newer generation premixed bioceramics have been introduced. These include NeoPUTTY®, Total Fill® BC UNIVERSAL RRM™, and Bio-C® Repair, each exhibiting unique compositional and functional properties designed to enhance clinical performance and ease of use.

Despite promising individual results, no clinical study has yet compared these three materials within the context of pulpotomy in immature permanent molars with irreversible pulpitis. This randomized clinical trial aims to fill this gap by evaluating their clinical and radiographic outcomes over a 12-month period, to better guide material selection in vital pulp therapy.

ELIGIBILITY:
Inclusion Criteria:

* -Healthy patients (according to ASA classification) with noncontributory medical history.
* Patients aged between 7 and 11 years of age, with at least one immature permanent molar with deep caries, needing full pulpotomy.
* Cooperative pediatric patients (Frankl's behavioral rating scale).
* Restorable immature permanent molar with deep caries: caries involving the pulpal roof or where complete caries removal would likely result in pulpal exposure.
* Physiological mobility.
* Vital pulp (detected by clinical signs/symptoms) presenting symptoms classically indicative of irreversible pulpitis according to AAE diagnostic criteria : positive but heightened response to cold sensibility testing, presence of spontaneous pain.
* No clinical signs of pulp necrosis; absence of a sinus tract or swelling.
* Patients who agree to return for periodic examination (follow-up).
* Patients who are willing to sign the consent form (written informed consent).

Exclusion Criteria:

* -Medically compromised patients.
* Patients older than 11 years or younger than 7 years of age.
* Mature permanent molar.
* No signs and symptoms of irreversible pulpitis.
* No pulp exposure even after complete caries excavation.
* Clinical signs of pulp necrosis on the tooth to be treated, such as insufficient bleeding or no bleeding after pulp exposure.
* Uncontrollable pulp hemorrhage (more than 10 minutes of hemostasis).
* Teeth previously endodontically treated.
* Teeth with pathological root resorption.
* Impossibility to place a rubber dam.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-02-27 (Estimated); Study Completion 2027-02-27 (Estimated)

PRIMARY OUTCOMES:
-Root formation and apical closure. | 12 months
  Continued root formation and apical closure will be assessed using standardized periapical radiographs of the treated immature permanent molars and classified according to Cvek's stages of root development. Radiographic evaluation will be performed by a calibrated examiner. Progression in root development will be determined by changes in root length and apical foramen morphology compared with baseline.
  Cvek's classification includes five radiographic stages of root development:
  Stage I (A): < 1/2 root length
  Stage II (B): 1/2 root length
  Stage III (C): 2/3 root length
  Stage IV (D): Nearly complete root length with wide open apical foramen
  Stage V (E): Complete root development with closed apical foramen
-Postoperative pain. -Percussion and/or palpation pain. | 12 months
  Pain response will be recorded as a binary outcome (Yes/No) based on the patient's subjective report during standardized clinical examination. The assessment will be performed by a calibrated examiner using gentle vertical percussion and periapical palpation according to routine endodontic diagnostic procedures.
  Measurement Tool
  Clinical percussion test
  Clinical palpation test
  Patient-reported pain response during examination (verbal report) Postoperative pain assessed using a Visual Analog Scale (VAS) ranging from 0 (no pain) to 10 (worst pain imaginable), recorded by the patient.

OTHER OUTCOMES:
-Presence of periapical lesion. | 12 months
  Presence of periapical lesion assessed on standardized periapical radiographs using the Periapical Index (PAI); lesions defined as a PAI score ≥ 3.

CONTACTS AND LOCATIONS:
Locations (1):
- Universite Saint Joseph de Beyrouth, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2026-01-09): https://cdn.clinicaltrials.gov/large-docs/46/NCT07350746/Prot_SAP_ICF_000.pdf